CLINICAL TRIAL: NCT00055432
Title: Gemzar (Gemcitabine) and Alimta (Pemetrexed) in the Treatment of Patients With Recurrent Platinum-Sensitive and Platinum-Resistant Ovarian or Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 7127; H3E-US-JMFU
Record Dates: First submitted 2003-03-03; First posted 2003-03-04 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Ovarian Cancer; Peritoneal Cancer
Keywords: recurrent ovarian cancer; platinum-resistant; platinum-sensitive; folate receptor antagonist
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Gemcitabine; Pemetrexed

INTERVENTIONS:
Drug: Gemzar and Alimta

SUMMARY:
This study hopes to evaluate whether the combination of Gemzar plus Alimta will have any beneficial effects for patients with recurrent platinum-sensitive or platinum-resistant ovarian or peritoneal cancer. Treatments are weekly for two weeks, with the 3rd week off and will be repeated every 21 days. Side effects and the overall safety of the treatment will also be monitored and evaluated. In addition, a Quality of Life questionnaire is part of this study to help measure patient perceived benefits or drawbacks to this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have disease that can be measured.
* Patients must meet criteria for either platinum-resistant or platinum-sensitive ovarian or peritoneal cancer.
* Patients may only have had one prior platinum-based chemotherapy regimen.
* Patients must be willing and able to stop all aspirin and NSAID medications immediately before and for a time after each treatment cycle (approx. 5-8 days)
* Patients must have normal kidney function.

Exclusion Criteria:

* Patients may not have a Low Malignant Potential or Borderline Ovarian Tumor.
* Patients may not have received pelvic or abdominal radiotherapy.
* Patients must not have evidence of or received treatment for another cancer within the last 5 years.
* Patients must not have been diagnosed with a heart attack in the last 6 months.
* Patients who are unwilling or unable to take folic acid tablets, vitamin B12 injections or dexamethasone tablets.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Atlanta, Georgia, United States